CLINICAL TRIAL: NCT03733431
Title: Non-invasive TRanscutaneous Cervical Vagus Nerve Stimulation as a Treatment for Acute Stroke; Safety and Feasibility Study
Acronym: TR-VENUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish Stroke Research and Clinical Trials Network (Network)
Collaborators: Turkish Neurological Society (Unknown); ElectroCore INC (Industry)
Responsible Party: Principal Investigator, Ethem Murat Arsava, Professor of Neurology, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TR-VENUS
Record Dates: First submitted 2018-11-03; First posted 2018-11-07 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Stroke; Stroke, Hemorrhagic
Keywords: vagal nerve stimulation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Standard dose vagal stimulation (Active Comparator): A total of 7 consecutive 2-minute trains at every 10 minutes for one hour (n=20)
  Interventions: Device: Gammacore device
- High dose vagal stimulation (Active Comparator): A total of 7 consecutive 2-minute trains applied at every 10 minutes for one hour that is followed by an additional 7 consecutive 2-minute trains interspersed at every 10 minutes applied 3 hours after completion of the initial scheme (n=20)
  Interventions: Device: Gammacore device
- Sham stimulation (Sham Comparator): A total of 7 consecutive 2-minute trains at every 10 minutes for one hour (n=20)
  Interventions: Device: Gammacore sham device

INTERVENTIONS:
Device: Gammacore device — Transcutaneous stimulation of vagus nerve with the device positioned below the mandibular angle, medial to the sternocleidomastoid muscle and lateral to the larynx.
  Arms: High dose vagal stimulation; Standard dose vagal stimulation
Device: Gammacore sham device — Sham device which does not deliver electrical stimulation, but instead, produces a buzzing sound will be placed along the lateral border of the sternocleidomastoid muscle in order to avoid mechanical stimulation of the vagus nerve in the carotid triangle.
  Arms: Sham stimulation

SUMMARY:
This study aims to determine safety and feasibility of non-invasive transcutaneous cervical Vagus nerve stimulation (nVNS) when delivered promptly after clinical diagnosis of acute stroke. Vagus nerve stimulation will be performed via GammaCore® device. A total of 60 patients will be randomized to each of 3 different groups; 'standard dose' vagal stimulation, 'high dose' vagal stimulation, and 'sham stimulation' (1:1:1 ratio). Adverse device events, serious adverse device events, and feasibility of vagal nerve stimulation at the setting of acute stroke will be evaluated. The study will be performed in a multi-center fashion among stroke centers within TurkStrokeNet Network.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are older than 18 years old who have been admitted to neurological intensive care or stroke units with ischemic or hemorrhagic stroke
* Patients with symptom onset time within 6 hours or with unknown time of onset and no evidence of acute ischemia on fluid attenuation inversion recovery (FLAIR) imaging
* Patients who have given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Patients who have a pre-stroke disability ≥ 2 according to the modified Rankin Score
* Patients who have a NIH Stroke Scale/Score (NIHSS) ≤ 4 or ≥30
* Patients who have a NIHSS item 1a ≥2
* Patients who have experienced early dramatic neurological improvement (NIHSS score improvement ≥8) prior to study randomization suggesting resolution of signs/symptoms of stroke
* Patients with classical lacunar syndrome
* Patients who have local infection, rash or space occupying lesion at the stimulation site
* Patients with a prior injury to the vagus nerve (cervical vagotomy)
* Patients with conditions that make the positioning of the device not possible such as tonic head deviation or involuntary movements of the head and neck
* Patients using medications that can interfere with central neurotransmitter mechanisms potentially involved in the central vagal pathway (complete list is provided below under concomitant medications)
* Patients with known severe (>90% stenosis) bilateral carotid artery disease
* Patients with known carotid hypersensitivity
* Patients who had undergone bilateral carotid endarterectomy or neck surgery involving the region of carotid triangle
* Patients who have low blood pressure (Baseline SBP≤100 mmHg or DBP≤60 mmHg)
* Patients who have slow heart rate (Baseline HR≤60/min)
* Patients who have high blood pressure (SBP>220 mmHg or DBP>130 mmHg) despite initial line of treatment
* Patients who have been involved in any investigational study within the previous 90 days
* Patients who have any terminal illness such that the patient would not be expected to survive more than 90 days
* Pregnant women
* Patients with severe hypoglycemia at admission (<60 mg/dl)
* Patient experiencing seizures
* Patients with baseline ECG showing first-degree AV block; second- or third-degree atrio-ventricular block with no pacemaker/ICD in place; or ventricular tachycardia/fibrillation
* Patients with digitalis toxicity
* Patients who are suspected to have an acute coronary syndrome after clinical evaluations (Clinical, ECG, or any related biomarker)
* Patients who are scheduled to have an emergent carotid artery angioplasty stenting or endarterectomy
* Patients implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
* Patients implanted with metal cervical spine hardware or having a metallic implant near the GammaCore stimulation site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular effects, clinical worsening or death (primary safety measure) | 24 hours
  any of the following:
  * severe bradycardia (HR ≤50/min) during treatment application
  * significant decrease in arterial blood pressure (≥20 mmHg decrease in mean arterial blood pressure) during treatment application
  * neurological worsening (progression of neurologic deficit as shown by ≥ 4 points increase in NIH Stroke Scale Score) within 24 hours
  * death within 24 hours

OTHER OUTCOMES:
Proportion of treatment eligible patients (feasibility measure 1) | 6 hours
  Proportion of eligible patients in whom nVNS can be started within the first 6 hours.
Proportion of patients completing all pre-specified treatment doses (feasibility measure 2) | 12 hours
  Proportion of enrolled patients who receive all the pre-specified treatment doses per protocol.
Stroke onset to treatment time (feasibility measure 3) | 6 hours
  Time from stroke onset to administration of the first dose of nVNS.
Early neurological outcome (efficacy measure 1) | 24 hours
  Proportion of patients with NIHSS score≤4 or improvement of baseline NIHSS score ≥8 at 24 hours
Early tissue outcome (efficacy measure 2) | 24 hours
  Delta infarct volume between baseline DWI and 24 hr MRI.
Local reaction at application site (secondary safety measure 1) | 12 hours
  Local irritation or skin reaction during treatment application
Acute coronary syndrome (secondary safety measure 2) | 24 hours
  Acute coronary syndrome
Symptomatic intracerebral hemorrhage (secondary safety measure 3) | 24 hours
  Symptomatic intracerebral hemorrhage: ≥ 4 points increase in NIH Stroke Scale Score (NIHSS) together with a PH2 (parenchymal hematoma-2) type intracerebral hemorrhage
Death, clinical worsening, and acute coronary syndrome (secondary safety measure 4) | 24 hours
  Combined outcome of death, clinical worsening, and acute coronary syndrome
New ischemic lesion or increase in hemorrhage (secondary safety measure 5) | 24 hours
  New, spatially distinct remote ischemic lesion outside the arterial territory of the index lesion on MRI at 24 hours or greater than 30% increase in hemorrhage volume from baseline CT to 24 hour MRI in the subset with intracerebral hemorrhage
Serious adverse device event (SADE) rate (secondary safety measure 6) | 24 hours
  Serious adverse device event (SADE) rate at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ethem M Arsava, MD, Principal Investigator — Hacettepe University; Mehmet A Topcuoglu, MD, Principal Investigator — Hacettepe University; Hakan Ay, MD, Study Chair — Massachusetts General Hospital, Harvard University
Locations (8):
- Turkey (Türkiye) (8):
  - Ankara University Faculty of Medicine, Ankara
  - Gazi University Faculty Of Medicine, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Akdeniz University, Antalya
  - Eskişehir Osmangazi Faculty of Medicine, Eskişehir
  - Necmettin Erbakan University, Konya
  - Selcuk University, Konya
  - Ondokuz Mayıs University Faculty of Medicine, Samsun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arsava EM, Topcuoglu MA, Ay I, Ozdemir AO, Gungor IL, Togay Isikay C, Nazliel B, Kozak HH, Ozturk S, Yilmaz IA, Dora B, Ay H; TR-VENUS investigators. Assessment of safety and feasibility of non-invasive vagus nerve stimulation for treatment of acute stroke. Brain Stimul. 2022 Nov-Dec;15(6):1467-1474. doi: 10.1016/j.brs.2022.10.012. Epub 2022 Nov 7. PMID 36356829